CLINICAL TRIAL: NCT06384989
Title: Phase II - Safety-Enhancing Motor Vehicle Child Safety Seat
Brief Title: Safety-Enhancing Motor Vehicle Child Safety Seat
Status: Completed | Type: Observational
Sponsor: Minnesota HealthSolutions (Industry)
Responsible Party: Principal Investigator, Julie Mansfield, Research Assistant Professor, Minnesota HealthSolutions
Other Study IDs: MinnesotaHealthSolutions_LL
Record Dates: First submitted 2024-04-18; First posted 2024-04-25 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Motor Vehicle Injury; Safety Issues
Keywords: child restraint system
MeSH Terms: interventions — Child Restraint Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Child restraint system with load leg feature — The primary objective is to assess the usability of the load leg design for caregivers who must install the child safety seat into a vehicle. The specific aims are to quantify any errors committed by the participants while installing the car seat (especially related to the use of the load leg) and to assess participants' opinions on the car seat's load leg design.

SUMMARY:
This study aims to assess the usability of a load leg design for caregivers who must install the child safety seat into a vehicle. The specific aims are to quantify any errors committed by the participants while installing the car seat and to assess participants' opinions on the car seat's load leg design.

DETAILED DESCRIPTION:
A descriptive study will be conducted to determine whether human subjects are able to install the new feature of the prototype car seat correctly. Participants will be presented with the prototype car seat and a set of basic written instructions and labels to guide their installations. The percentage of participants who use the new feature and use it correctly will be reported. Any installation errors on other parts of the child seat (seat belt, lower anchors, top tether) will also be reported.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Be a care provider to a child who is up to 4 years of age
* Have installed a child safety seat in the last 2 years
* Able to lift and install a child safety seat into a vehicle
* English-speaking (because consent forms and explanation will be given in English)

Exclusion Criteria:

* Not meeting any of the above

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be recruited from the Central Ohio area. Adults who meet the above criteria will be enrolled. Efforts will be made to include both males and females, across a range of ages, as well as minorities, as these groups' experiences around child seats may vary.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-05-22 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Mansfield, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Data will be available upon request after publication of the results.

RESULTS

PARTICIPANT FLOW:
Groups:
- Single-group Study: All 50 participants were part of a single group. Their interactions with/installations of the prototype child seat with a load leg were observed.
Period: Overall Study
Arm/Group | Single-group Study
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single-group Study
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 37
  More than one race | 3
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Overall Correct Use of Load Leg
Description: Number of participants who correctly install the load leg independently, without needing any prompt to use it.
Time Frame: 1 study visit, an average of 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Single-group Study
Number analyzed (Participants) | 50
Participants | 18

2. Primary Outcome: Attempt to Use Load Leg Without Prompting
Description: Number of participants who noticed the load leg on their own, unfolded it from storage, and attempted to use it without being prompted by the researcher.
Time Frame: 1 study visit, an average of 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Single-group Study
Number analyzed (Participants) | 50
Participants | 27

3. Primary Outcome: Correct Load Leg Length
Description: Number of participants who set the load leg to the correct length, including those who needed prompted to use it
Time Frame: 1 study visit, an average of 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Single-group Study
Number analyzed (Participants) | 50
Participants | 35

4. Primary Outcome: Correct Load Leg Angle
Description: Number of participants who set the load leg to the correct angle, including those who needed prompted to use it.
Time Frame: 1 study visit, an average of 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Single-group Study
Number analyzed (Participants) | 50
Participants | 37

5. Secondary Outcome: Correct Understanding of Load Leg's Purpose
Description: The number of participants who correctly understood the purpose of the load leg by using words such as "security, safety, stability," etc. in their survey responses.
Time Frame: 1 study visit, an average of 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Single-group Study
Number analyzed (Participants) | 50
Participants | 48

6. Secondary Outcome: Participants Who Like Having the Load Leg
Description: Number of participants who overall reported that they would like having the load leg feature on a child seat.
Time Frame: 1 study visit, an average of 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Single-group Study
Number analyzed (Participants) | 50
Participants | 28

ADVERSE EVENTS:
Time Frame: During study tasks which took approximately 30 minutes to complete. The study involved minimal risk only. Participants installed a child seat into a vehicle, which is a typical task of adults and caregivers.
Arm/Group | Single-group Study
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT06384989/Prot_SAP_000.pdf